CLINICAL TRIAL: NCT06012474
Title: Effect Of Power Breath Device On Arterial Blood Gases And Diaphragmatic Excursion After Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Mahdy Hassan Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 012/004209
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inspiratory muscle training group (Experimental): 30 patients will receive inspiratory muscle training by Power breath device once daily for 7 days.
  Interventions: Other: Power breath plus; Other: Incrementing the training load
- diaphragmatic breathing exercise group (Active Comparator): 20 patients will receive program of diaphragmatic breathing exercise by incentive spirometer once daily for 7 days.
  Interventions: Other: Diaphragmatic breathing exercises

INTERVENTIONS:
Other: Power breath plus — Power breath plus use a variable load calibrated spring. It can be adjusted from the lowest load setting (17cmH2O) when training began and increased as the patient breathing muscles adapt and become stronger (maximum load setting 274cmH2O). Use a comfortable chair, preferably straight-back so that the spine is straight at all times during the exercise. patients will be instructed to exhale calmly, followed by a maximal forced inspiration to total lung capacity using a mouthpiece and a nasal clip as an aid to prevent air leaks and will ask to make 10 breaths for 3 sets once daily for 7 days with 2min rest between sets
  Arms: inspiratory muscle training group
Other: Incrementing the training load — The resistance will be increased incrementally, based on the rate of perceived exertion (RPE) scored by the patient on the modified Borg Scale. If the RPE is less than 5, the resistance of the inspiratory trainer will be increased incrementally by 2cmH2O. The resistance will not change if the level of perceived exertion is rated from 6 to 8, and the resistance will be decreased by 1 to 2 cmH2O if the level of perceived exertion is rated 9 or 10.
  Arms: inspiratory muscle training group
Other: Diaphragmatic breathing exercises — Training by using incentive spirometer:
  * Loosen any tight clothing, especially around neck.
  * Each patient will be instructed to sit upright with placing incentive spirometer at the same level of his mouth to promote optimal lung expansion while using the spirometer.
  * The patient will be instructed to exhale letting all the breath out.
  * patient will asked to close the lips around the mouthpiece of the spirometer.
  * patient will be instructed to inhale slowly, breathing in until unable to do any more, this would raise the balls to the top of the column.
  * patient will be asked to hold the breath as long as possible (at least five seconds) then exhale slowly.
  * Session will be in the form of 30 times in sets, each set consist of 5-6 repetitions with rest 1 minute between sets.
  * Intensity of exercise will be increased by increasing time of session, time of holding the breath and numbers of repetitions according to patient's status.
  Arms: diaphragmatic breathing exercise group

SUMMARY:
The aim of this study is to evaluate the effect of power breath device on arterial blood gases, diaphragmatic excursion and the 6 min walk test after cardiac valve surgery.

DETAILED DESCRIPTION:
No more studies have been done on the effect of IMT by power breath on valvular surgery, So, this study will see the effect of power breath device on arterial blood gases, diaphragmatic excursion and six minute walk test after valve surgery to know enhanced recovery protocols in valvular surgery that accelerate the functional recovery, minimize the length of the hospital stay and decrease cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with valve surgery (valve replacement or repair with median sternotomy procedure).
* Age between 25 to 35 years old.
* BMI is between 18.5 to 24.5 kg/m2.

Exclusion Criteria:

The participants will be excluded if they meet one of the following criteria:

* Uncontrolled hypertension (systolic blood pressure>230 mm Hg and diastolic blood pressure>120 mm Hg)
* Patients with coronary artery disease or heart failure.
* Need for mechanical ventilation for >24 h or reintubation.
* Renal and hepatic disorders.
* Infected or unstable sternum.
* patient with pneumothorax after surgery.
* Metabolic disorders.
* Pregnant woman.
* Lactating mother.
* Smokers
* Stroke patient

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in diaphragmatic excursion | within 24 hours after 1 week of intervention
  By using Ultrasonography (Aloka prosound 4000, made in Japan) that will be used to assess diaphragmatic excursion. Diaphragmatic excursion is measured 3 times :at baseline before surgical intervention, second day after surgery (before the training program) and after 7 days of training program for all patient in the two groups. Diaphragmatic excursion was measured during deep breathing while the patient in semi-recumbent position on a comfortable bed using ultrasonography.
Assessing the change in Arterial Blood gases | within 24 hours after 1 week of intervention
  Arterial blood gases are measured at baseline before surgical intervention, second day after surgery (before the training program) and after 7 days of training program for all patient in the two groups and can be obtained by direct arterial puncture most usually at the wrist (radial artery), femoral and brachial artery. An arterial blood sample (2 to 3 ml) will be collected.
Assessing the change in capacity to perform daily activities | within 24 hours after 1 week of intervention
  by using the The 6-min walk test (6MWT) is a submaximal functional test indicative of the capacity to perform daily activities, patients will be asked to walk along a 30-m, flat and straight hospital corridor. Encouragement will be offered every minute, so that subjects will walk as far as possible. Symptom-limited interruptions (dyspnea, skeletal muscle pain, angina, dizziness) will allowed, though patients will be invited to resume walking as soon as possible. Most tests will be supervised by a physical therapist. Distance will be recorded in meters. Subjective dyspnea will quantified according to Borg Scale, ranging from 0 (no dyspnea) to 10 (severe dyspnea).

CONTACTS AND LOCATIONS:
Overall Officials: Hend Mahdy, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No